CLINICAL TRIAL: NCT06441500
Title: Child Oral Health Pilot Programme - SmilebrightRO
Brief Title: Oral Health and Dental Caries Prevention Intervention for Children in Romania
Acronym: Smilebright
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Grigore T. Popa University of Medicine and Pharmacy (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other); George Emil Palade University of Medicine, Pharmacy, Sciences and Technology of Targu Mures (Other); University of Medicine and Pharmacy Craiova (Other)
Responsible Party: Principal Investigator, Basaraba Gabriela Lavinia, Head of grant department, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18688/16.10.2023
Record Dates: First submitted 2024-04-19; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries; Early Childhood Caries; Quality of Life
Keywords: dental caries; quality of life; diet; socio-economic status; county development index
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kindergarten children (Experimental): Children aged 3-5 years, enrolled in kindergartens. The pathfinder sampling technique has been used to obtain a representative sample. As suggested by the WHO, this survey design is suitable for collection of data for planning purposes and monitoring of oral health programmes in all countries regardless of the level of disease, availability of resources or complexity of care. Clinical examinations will be performed using ICDAS criteria by calibrated medical staff from each partner university. Caries incidence rate will be calculated on each tooth as the unit of analysis and evaluated using a multi-step approach: net increment for caries severity using ICDAS calculated at each follow-up examinations; Events defined as a new lesion or as the sum of the Δ-caries changes of status recorded at the baseline, at interim, and at the last examination. The number of events will be appraised by subtracting the number of caries-free teeth at last examination from those at baseline.
  Interventions: Other: Daily tooth brushing programme

INTERVENTIONS:
Other: Daily tooth brushing programme — Implementing the toothpaste/toothbrushing scheme involving free daily toothbrushing to every 3 - 5-year old child attending nursery. Free distribution of toothpaste/toothbrush packs to every child every 3 months. Collection of routine monitoring data linked with national data sets from the previous survey regarding caries prevalence and risk factors.2.Monitor caries activity - net caries increment for initial, moderate, and extensive caries severity.

SUMMARY:
During 2019-2020, the National Oral Health Survey evaluated a significant sample of children aged 5, 6 and 12 years, gathering baseline data on oral health. Data was used to estimate the distribution and severity of dental caries, the need for community-oriented disease prevention and health promotion, and the nature of oral health intervention(s) required. The survey also established how younger age groups can be reached and evaluated. Only 14% of 6 years old children have dmft 0 and the SiC index of the same sample is 9.83. High prevalence of tooth decay with high severity scores, significant inequalities in oral health and poor use and access to services showed the need for a child oral health programme.

The originality of the project lies in the vision of using fluoridated toothpaste not only as a means of preventing new carious lesions but also in the therapeutic effect of fluoridated toothpaste, which the study set out to evaluate. This programme could represent an example of good practice for the countries in our region, starting from downstream oral health interventions, such as clinical prevention and oral health promotion, and developing towards upstream interventions.

The aim of the project is to improve oral health and reduce inequalities both in dental health and access to dental services by shifting the balance of care towards preventive care.

The programme is structured on three levels:

1. Specific training for dental hygienists to deliver oral health promotion to children and nursery educators, focus on tailoring key messages outlined in the care pathway and practical preparation for delivering interventions in nurseries.
2. A toothpaste/toothbrushing scheme involving free daily toothbrushing to every 3 and 4-year old child attending nursery.
3. Provision of clinical prevention activities delivered by dental hygienists for children attending nurseries.

The evaluation of the programme consolidates and builds upon previous evaluation work of the National Oral Health Survey for children. Due to the fact that it is a pilot programme aiming to be further implemented at national level, an evolving model of evaluation is appropriate. This allows the evaluation to be responsive to issues emerging from its implementation and develops the programme as a result of the evaluation findings.

DETAILED DESCRIPTION:
Until recently, Romania has lacked baseline data regarding the oral health status of children. A previous study by Petersen et al. was conducted in the 1990s covering only five major cities and without taking into account rural areas. Some local papers described a high caries prevalence. Only one longitudinal study assesses caries trends in Romanian schoolchildren. A contemporary assessment was therefore mandatory in order to advance scientific understanding and allow for the development of adequate public health policies. During 2019-2020, the National Oral Health Survey financed by The Borrow Foundation, evaluated a significant sample of children aged 5, 6 and 12 years, gathering baseline data on oral health according to the WHO guidelines. The data was used to estimate the distribution and severity of dental caries, the need for community-oriented disease prevention and health promotion, and the nature and urgency of the oral health intervention(s) required. The survey also established how younger age groups can be reached and evaluated. Unpublished data show that only 14% of 6 years old children have dmft 0 and the SiC index of the same sample is 9.83. High prevalence of tooth decay with high severity scores, significant inequalities in oral health and poor use and access to services showed the need for a child oral health programme.

The main objectives of the program are to:

1. Reorient the traditional curative approach, which is basically pathogenic, and move towards a preventive promotional approach
2. Strengthen cross-sectoral collaboration across key settings, such as schools, communities and workplaces to promote habits and healthy lifestyles, integrating teachers and the family;
3. Raising the priority accorded to the prevention and control of oral diseases in regional and national agendas and development goals, through strengthened cooperation and advocacy.

The programme is designed to deliver additional clinical prevention activities through dental hygienists, aimed at children aged three years and above attending priority nursery establishments in order to improve oral health of young children, and complemented the established national toothpaste/toothbrushing scheme.

The programme will be implemented for a period of 24 months, under guidance from the WHO Collaborative Centre for Epidemiology and Community Dentistry Milan, Italy. Consent from the national and regional authorities will be obtained, nurseries will be informed and the informed consent of the parents will be asked. The total sample size will be calculated according to the WHO guidelines using a stratified sampling technique for examination sites in Bucharest, Timisoara, Cluj-Napoca, Craiova, Iasi, Targu Mures and the surrounding geographical area. The programme will be conducted in collaboration with the Universities of Medicine in the capital and the cities mentioned above, under supervision of the university staff. Data collection points will be 4 kindergartens in the Capital or metropolitan areas, 2 kindergartens in each of 2 large cities, and 1 kindergarten in each 4 villages from different geographic areas.

The programme fits in the Oral Health Resolution of the Seventy-fourth World Health Assembly (WHA 74.5 - 31.05.2021) aiming at:

* understanding and addressing the key risk factors for poor oral health and associated burden of disease;
* fostering the integration of oral health within their national policies, including through the promotion of articulated interministerial and intersectoral work;
* reorienting the traditional curative approach, which is basically pathogenic, and move towards a preventive promotional approach with risk identification for timely, comprehensive and inclusive care;
* strengthen cross-sectoral collaboration across key settings, such as schools, communities and workplaces to promote habits and healthy lifestyles, integrating teachers and the family; The study design takes into consideration all principles stated in the WHO Implementation Manual "Ending childhood caries": Early diagnosis of caries lesions through clinical examinations in the nurseries, control of risk factors trough the evaluation of oral health related knowledge and behaviours and health education, arresting caries through the application of fluoride varnishes, developing primary care teams by introducing a new workforce - dental hygienists, building a framework to integrate prevention and control of dental caries into general health interventions.

The project will be implemented in collaboration with the universities of Medicine and Pharmacy in the country to ensure a homogeneous distribution of evaluation sites. Selection of nurseries will be done according to the pathfinder sampling technique. This survey design is suitable for collection of data for planning purposes and monitoring of oral health programmes in all countries regardless of the level of disease, availability of resources or complexity of care. The principles of the sampling techniques are the following:

* The study supposes a sample of 460 children;
* There are 6 universities involved in data collection;
* Data will be collected from 3 types of residential areas: metropolitan areas (180 evaluations); big cities (180 evaluations), rural areas (100 evaluations);
* In metropolitan areas and big cities, 25 children have to be evaluated in the same kindergarten.
* In rural areas, more than one kindergarten can be evaluated until the desired number of evaluations is obtained for the specific region. This principle has been added because kindergarten is not mandatory in Romania and the number of children enrolled in kindergarten in rural areas is quite low in some regions of the country.

Distribution of data collection points:

* University of Medicine and Pharmacy Bucharest will provide:

  * 25 evaluations in one kindergarten in Bucharest;
  * 25 evaluations in rural areas of surrounding counties
* University of Medicine and Pharmacy Cluj will provide:

  * 25 evaluations in one kindergarten in Cluj Napoca;
  * 25 evaluations in rural areas of surrounding counties;
* University of Medicine and Pharmacy Craiova will provide:

  * 25 evaluations in 2 kindergartens in Drobeta-Turnu Severin;
  * 25 in rural areas of surrounding counties;
* University of Medicine and Pharmacy Iași will provide:

  * 25 evaluations in 2 kindergartens in Iași (2 X 25 = 50);
  * 25 in rural areas of surrounding counties;
* University of Medicine and Pharmacy Targu Mures will provide:

  * 25 evaluations in one kindergarten in Targu Mures;
  * 25 evaluations Miercurea Ciuc;
* University of Medicine and Pharmacy Timișoara will provide:

  * 25 evaluations in one kindergarten in Timișoara;
  * 25 evaluations in 2 kindergartens in Arad; According to the WHO STEPS approach, results from the first two steps - self-evaluation and collection of clinical data will be used to plan and evaluate further health interventions.

Volunteer dental hygienists students will be trained deliver oral health promotion to nursery educators and oral health promotion activities for children, focusing on tailoring of key messages to the specific age and on practical preparation for delivering interventions in the nurseries along with implementing the toothpaste/tooth brushing scheme involving free daily tooth brushing to every 3 and 4-year old child attending nursery.

The evaluation of the programme consolidates and builds upon previous evaluation work of the National Oral Health Survey for children. Due to the fact that it is a pilot programme aiming to be further implemented at national level, an evolving model of evaluation is appropriate. This allows the evaluation to be responsive to issues emerging from its implementation and develops the programme as a result of the evaluation findings.

Methods used in the evaluation have to be formative - to adapt the programme, and summative - to assess its impact. Evaluation activity includes the collection of routine monitoring data linked with national data sets from the previous survey, assessment of the programme's impact at different time-intervals, and assessment of economical outcomes.

One of the outcomes will be to assess oral health practices of children using the previously designed questionnaire from the National Oral Health Survey, meaning to describe oral health behaviour of the evaluated children in correlation to the 'County Development Index', residential area, type of residence, characteristics of the parents (education, working status) and characteristics of the child (age, gender). The County Developmental Index is a sociological index that combines county-level variables: education stock, life expectancy at birth, medium age of adult population, average living space, number of private cars to 1000 inhabitants, and average household gas consumption. Another secondary outcome will establish correlations between the levels of oral health knowledge and clinically detected oral health status and assess the impact of the intervention on the oral and general health status.

Monitoring the quality of the intervention delivered by dental hygienist students will assure the necessary information to change/adapt their education to the necessary actions.

Short term outcomes will be:

* Increased level of knowledge and improved oral health behaviours for children in this age group
* Reduced risk of new carious lesions and progression of existing lesions
* Improved skills of a new profession - dental hygienists and shift of workforce
* Improvement of the existing data base and implementation of a monitoring activity at national level

Other potential outcomes:

* Improved knowledge and behaviour within the families which might lead to an improvement of oral but also general health status
* Reduced inequalities in oral health care
* Reduced treatment needs and therefore reduced costs for dental treatment The research team proposed to incorporate sustainability into the process taking into account the fact that health interventions often include a number of unquantifiable variables, which add a layer of complexity in terms of environmental appraisals. The discrepancy between the existence of evidence-based health promotion interventions and their use in practice is present in almost all medical fields, but has been widely recognized as a challenge in dentistry. Clearly, the traditional modes of spreading information through scientific publication channels and passive instruction are not sufficient to reliably initiate and sustain new practices. In order to move evidence-based approaches into practice, more careful examinations of methods to introduce and sustain effective oral health practices are needed. For this project we suggested a framework multi-staged approach. This resource is designed to interweave with the many other point of the project that have been developed to guide oral health professionals and dental organizations.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3-5 years attending public nurseries in Romania

Exclusion Criteria:

* enamel fluorosis
* enamel developmental defects
* incapacity to perform tooth brushing by themselves

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic baseline data on caries prevalence | 3 months
  Prevalence will be determined for the specific age group after primary examination using ICDAS criteria after calibration. Children will be examined in a seated position, using a dental mirror and a probe, without air-drying. Thus, ICDAS codes 1 and 2 will be counted together as "A".
  To evaluate the outcomes, a statistical analysis will be performed. All the data will be input into a spreadsheet (Microsoft Excel 2021 for Mac, version 16.4.8).The total number of existing caries will serve for the calculation of the dmft index (decayed-missing-filled teeth index) and the SiC index (Significant caries index).
Epidemiologic baseline data on caries severity | 3 months
  Clinical examinations will be performed using ICDAS criteria by calibrated medical staff from each partner university after calibration. Children will be examined in a seated position, using a dental mirror and a probe, without air-drying. Thus, ICDAS codes 1 and 2 will be counted together as "A". Statistical analysis will be performed after inputing the data into a sheet (Microsoft Excel 2021 for Mac, version 16.4.8). Severity will be determined for the specific age group after primary examination using ICDAS criteria. ICDAS codes of 0 represent sound teeth, codes of 1 and 2 represent initial reversible caries lesions, only affecting the enamel, codes of 3 represent initial microcavitation of the enamel, codes of 4 represent moderate carious lesions and codes of 5 and 6 represent extended lesions.
Epidemiologic baseline self assessment data | 3 months
  Self-assessment of oral health behaviours of children will be done using the previously designed questionnaire from the National Oral Health Survey. The working tool consists of 15 items that make up the two types of behaviour (prevention and diet), and family characteristics (parent's level of education, working status). Behaviours will be correlated with clinical indices that will help us to delimit the existence or lack of certain significant differences among children. For a better understanding of the risk factors the evaluation relates to specific elements of the child (gender, age, parental education, residence), and elements related to the objective living conditions (county development index, residence, etc.). Statistical analysis using Poisson regression will correlate data obtained from self assessment with clinical outcomes expressed by the dmft index.
Monitor caries activity | 18 months
  Follow-up data regarding changes in caries status: new lesions appearing or existing caries status changes at interim and last examination. Caries incidence rate will be calculated on each tooth as the unit of analysis and evaluated using a multi-step approach:
  A - The net caries increment for initial, moderate, and extensive caries severity using ICDAS (Δ-initial, Δ- moderate, and Δ- extensive) will be calculated at each follow-up examinations; B - Events will be defined as a tooth getting a lesion or as the sum of the Δ-caries changes of status recorded at the baseline examination, at interim, and at the last examination. The number of events will be appraised by subtracting the number of caries-free teeth at last examination from those at baseline.
  The non-parametric Mann-Whitney U test will be applied to assess the differences across mean number of events between groups.
Efficacy of the treatment | 18 months
  The efficacy of the treatment will be assessed for those who fully followed the protocol (per-protocol subjects) by calculating the reduction in risk ratio (RR) and the related number needed to treat (NNT) value. An event is defined as the change of status at tooth level, i.e. the development of a new lesion or the progression of an existing lesion to a more severe stage.
  Cox Proportional Hazards models will be run to assess the factors associated with caries change of status. Estimates will be reported in the hazard ratio (HR) and their respective 95% confidence interval (95%CI). For all statistical analyses, the statistical significance will be set at α=0.05

SECONDARY OUTCOMES:
Daily tooth brushing pattern | 12 months
  Create a daily tooth brushing pattern in nurseries, with a particular focus on high risk communities
  * Habituation of daily tooth brushing in children
  * Skills in performing tooth brushing
Qualitative evaluation of the preventive activities in nurseries | 12 months
  Qualitative assessment of advantageds and barriers regarding the number of children who benefit from preventive measures will be done by means of interviews with the involved nursery staff
Qualitative evaluation of oral health promotion activities | 12 months
  Qualitative assessment of advantageds and barriers regarding the number of children who benefit from preventive measures will be done by means of interviews with the involved dental hygienists

CONTACTS AND LOCATIONS:
Overall Officials: Ruxandra Sava-Rosianu, Study Director — Victor Babes University if Medicine and Pharmacy Timisoara Romania
Locations (5):
- Romania (5):
  - University of Medicine and Pharmacy Cluj-Napoca, Cluj-Napoca, Cluj
  - University of Medicine and Pharmacy Craiova, Craiova, Dolj
  - County School Inspectorate Iasi, Iași, Iaşi
  - University of Medicine and Pharmacy Targu Mures, Târgu Mureş, Mureș County
  - University of Medicine and Pharmacy Bucharest, Bucharest

IPD SHARING:
Plan to Share IPD: No